CLINICAL TRIAL: NCT06161766
Title: Evaluation of the Natural History of Combined Hepatorenal Syndrome in Patients With Signs of Chronic Renal Disease
Brief Title: Terlipressin in Combined Hepatorenal Syndrome in Patients With Signs of Chronic Renal Disease
Acronym: Terli-CKD
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Collaborators: Jena University Hospital (Other); Johannes Gutenberg University Mainz (Other); University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dominik Bettinger, Deputy Principal Investigator, University Hospital Freiburg
Other Study IDs: Terli-CKD
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Liver Cirrhosis; Hepato-Renal Syndrome; Chronic Kidney Diseases
MeSH Terms: conditions — Liver Cirrhosis; Hepatorenal Syndrome; Renal Insufficiency, Chronic | interventions — Terlipressin; Albumins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with HRS-AKI or HRS-AKI-like syndrome and chronic kidney disease: Patients with clinical suspicion of HRS-AKI or HRS-AKI-like syndrome in case of previously diagnosed chronic kidney disease (CKD) who who receive vasoactive treatment for the management of HRS, as defined by the administration of terlipressin or noradrenalin plus albumin.
  Interventions: Drug: terlipressin or noradrenalin plus albumin

INTERVENTIONS:
Drug: terlipressin or noradrenalin plus albumin — Patients with clinical suspicion of HRS-AKI or HRS-AKI-like syndrome in case of previously diagnosed CKD who had received vasoactive treatment for the management of HRS, as defined by the administration of terlipressin or noradrenalin plus albumin.

SUMMARY:
The aim of this retrospective study is to evaluate the treatment response to terlipressin and albumin in patients with suspicion of HRS-AKI and signs of chronic parenchymal kidney disease (HRS-AKI-like syndrome) compared to patients without signs of chronic parenchymal kidney disease (HRS-AKI).

DETAILED DESCRIPTION:
Liver cirrhosis is a major cause of global health burden, accounting for 31 million disability adjusted life years and 1 million deaths worldwide in 2010. In the natural history of liver disease, there are two clearly distinct clinical phases. During the compensated phase, patients remain asymptomatic or oligosymptomatic. Although these patients may exhibit signs of cirrhosis, such as varices, spider naevi, or abnormalities in blood tests, they do not experience overt symptoms of the disease. The median survival rate for these patients is approximately 15 years 2. During the course of liver cirrhosis, patients may develop ascites, variceal bleeding or hepatic encephalopathy, which marks the transition to the decompensated phase of the disease. Thus, decompensation is associated with a significant reduction in survival, with a median of approximately 2 years, and ascites is the most frequent decompensating event. Clinically significant portal hypertension, as determined by the hepatic venous pressure gradient, is a main driver for the development of decompensation. In the decompensated phase, one can differentiate between patients who have a sole event as a decompensating event (typically ascites or variceal bleeding) and those who develop more than one decompensating event (further decompensation). These patients are at risk of dying due to their liver disease.

Hepatorenal syndrome refers to a "functional" renal dysfunction that occurs in patients with cirrhosis and ascites due to reduced renal perfusion secondary to hemodynamic alterations in the arterial circulation and activation of endogenous vasoactive system. Traditionally, one distinguished between hepatorenal syndrome type 1, which was a rapidly progressive renal failure (increase of serum creatinine (SCr) to greater than 2.5 mg/dL within two weeks) or hepatorenal syndrome type 2, which has a less rapid course, with a progressive increase of SCr to greater than 1.5 mg/dL. Typically, hepatorenal syndrome type 1 takes place in the context of an acute event, whereas hepatorenal syndrome type 2 takes place in end-stage refractory ascites.

In 2015, the International Club of Ascites (ICA) adopted a new classification of renal dysfunction in cirrhosis.

The decision was motivated by increasing evidence suggesting that serum creatinine could underestimate the real renal function in cirrhosis due to muscle wasting, increased tubular secretion of creatinine, increased volume of distribution potentially diluting creatinine and interference with bilirubin. Furthermore, the use of thresholds does not allow the flexibility that is required to confront a dynamic situation like hepatorenal syndrome type 1. To address these concerns, the ICA proposed to adopt criteria from The Kidney Disease: Improving Global Out-comes (KDIGO) guidelines, which define AKI as any of the following: 1) increase in SCr by ≥ 0.3 mg/dl (≥ 26.5 µmol/L) within 48 h; or 2) increase in SCr to ≥ 1.5x baseline, which is known or presumed to have occurred within the prior 7 days; or 3) urine volume < 0.5 ml/kg/h for 6 h. In the specific context of cirrhosis, the ICA proposed a modification by using only the first three KDIGO criteria, given the fact that urine output frequently does not properly reflect the renal function as patients with cirrhosis often are oliguric due to avid sodium retention or have a falsely high urine output due to the use of diuretics. Furthermore, ICA proposed that if a baseline value within the previous 7 days is unavailable, a SCr within the last 3 months before admission can be used.

According to the relative increase in creatinine, various stages of AKI can be identified. Noticeably, AKI can occur even when renal function remains within the given normal range. Within AKI Stage I, a differentiation can be made between individuals who achieve a peak over SCr ≥ 1.5 mg/dL (Stage Ib) and those who achieve a peak below this threshold (Stage Ia), the latter of which may have a similar survival as those without AKI and in whom the AKI is more frequently reversible.

AKI occurs in approximately 20 % of hospitalized patients with cirrhosis and is associated with higher mortality in patients with cirrhosis admitted to regular wards. Approximately 2/3 of AKI are due to renal hypoperfusion, which in turn can be divided into prerenal AKI (responsive to the administration of volume overload) or hepatorenal-AKI (HRS-AKI) (unresponsive to the administration of volume overload. HRS type 1 (now included in HRS-AKI) has a high mortality of almost 100 % when left untreated and is frequently part of multiorgan failure (acute on chronic liver failure). Among the etiologies of AKI in cirrhosis, hepatorenal AKI has the worst prognosis.

The diagnosis of HRS-AKI is based on ruling out other causes of AKI, mainly hypovolemia, ongoing infection, nephrotoxic medications, and intrinsic renal disease. Nevertheless, with the increasing incidence of MASLD (metabolic dysfunction associated steatotic liver disease) patients frequently have associated metabolic conditions (such as diabetes or arterial hypertension) which can lead to chronic renal injury and chronic kidney disease independent of liver cirrhosis and portal hypertension.

It's crucial to note that patients showing signs of parenchymal kidney disease at baseline cannot be classified as having HRS according to the current definition, but in occasion may have an AKI which follows the same pathophysiology as HRS (HRS-AKI-like syndrome).

Nevertheless, patients with HRS-AKI-like syndrome are regularly treated with vasoactive therapy, although this would be considered as off-label use in case of terlipressin.

Importantly, data regarding outcomes of this therapy in patients who do not fulfill the strict definition of hepatorenal syndrome are not available and are urgently needed.

The aim of the present study is to evaluate the treatment response to vasoactive therapy in patients who do not fulfill the criteria of hepatorenal syndrome due to the presence of signs of intrinsic nephropathy, but otherwise have a high suspicion of HRS-AKI (HRS-AKI-like syndrome). It is expected, that physicians considered the presence of a HRS-AKI-like syndrome as the dominating cause of AKI and a high proportion of patients were treated with terlipressin and albumin according to clinical practice. The secondary aims include the evaluation of 3-month, 6-month and 12-month survival rate, the improvement of renal function at different time-points (partial- or complete-response), the in-hospital mortality and duration of hospital stay as well as the need of renal replacement therapy, the need of LT during follow-up and the development of cirrhosis complications and acute-on-chronic liver failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis confirmed by histology or liver stiffness or with unequivocal signs in ultrasound, endoscopy and/or blood tests hospitalized between 1st of January 2018 and 31st of December 2022.
* Evidence of ascites due to portal hypertension
* Clinical suspicion of HRS-AKI or HRS-AKI-like syndrome (in case of previously diagnosed CKD)
* Pre-existing data on kidney function (SCr and eGFR) minimum 3 months prior to admission in a stable situation
* Dip stick urine test results (screening for proteinuria and hematuria) before initiation of AKI-treatment
* Vasoactive treatment for the management of HRS-AKI, as defined by the administration of terlipressin or noradrenalin plus albumin
* Age ≥ 18 years old

Exclusion Criteria:

* Uncontrolled shock
* Patients with cardiac cirrhosis as defined by the development of cirrhosis in a patient with chronic heart failure due to a primary cardiac disease (ischemic cardiomyopathy, hypertensive cardiomyopathy, etc.)
* Patients with hepatocellular carcinoma BCLC C or D
* Patients receiving renal replacement therapy at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed liver cirrhosis with ascites due to portal hypertension and 3) Clinical suspicion of HRS-AKI or HRS-AKI-like syndrome are included in this study. HRS-AKI-like syndrome is defined as typical features of HRS but wuth pre-existing chronic kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Complete response to treatment with vasoactive drugs and albumin at the end of treatment | Through study completion, an average of 12 months
  Complete response, as defined by a decrease of serum creatinine (SCr) to a value within 0.3 mg/dl (26.5 µmol/L) of the baseline value, at the end of vasoactive treatment.

SECONDARY OUTCOMES:
Complete response to treatment with vasoactive drugs and albumin during follow-up | Through study completion, an average of 12 months
  Complete response, as defined by a decrease of serum creatinine (SCr) to a value within 0.3 mg/dl (26.5 µmol/L) of the baseline value, at 3-months, 6-months and 12-months after treatment
Transplantation-free survival | Through study completion, an average of 12 months
  Transplantation-free survival is defined as survival without need for liver transplantation
Partial response, at the end of vasoactive treatment | Through study completion, an average of 12 months
  Partial response, at the end of vasoactive treatment defined as reduction of at least one AKI stage with decrease of serum creatinine to ≥ 0.3 mg/dl (26.5 µmol/L) of baseline value
In-hospital mortality | Through study completion, an average of 12 months
  In-hospital mortality is defined as death during index hospitalization
90-day survival | Within 90 days after beginning of hospitalization
  90-day survival is defined as survival assessed from beginning of hospitalization until 90 days after beginning of hospitalization
Length of in-hospital-stay | Through study completion, an average of 12 months
  Length of hospital stay is assessed from admission until discharge
Need for renal replacement therapy | Through study completion, an average of 12 months
  Beginning of renal replacement therapy
Recurrence of suspected HRS-AKI after treatment | Through study completion, an average of 12 months
  Recurrence of HRS-AKI
Complications of liver cirrhosis | Through study completion, an average of 12 months
  Development of complications of liver cirrhosis
Acute-on chronic liver failure (ACLF) | Through study completion, an average of 12 months
  Development of complications of ACLF

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ripoll, MD, Principal Investigator — University Hospital Jena; Dominik Bettinger, MD, Principal Investigator — University Hospital Freiburg
Locations (4):
- Germany (4):
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Medical center Jena, Jena
  - University Medical Center Mainz, Mainz
  - University Hospital Münster, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uschner FE, Schleicher EM, Passenberg M, Pohl J, Praktiknjo M, Volk AT, Karbannek H, Chang J, Grosse K, Rohrer C, Labenz C, Maasoumy B, Jamme P, von Widdern JC, Queck A, Trebicka J, Engelmann C, Rashidi-Alavijeh J, Bettinger D, Ripoll C; German Cirrhosis Study Group. Chronic Kidney Disease Does Not Influence Response to Terlipressin in Hepatorenal Syndrome-Acute Kidney Injury. Clin Gastroenterol Hepatol. 2025 Nov 19:S1542-3565(25)00989-9. doi: 10.1016/j.cgh.2025.11.006. Online ahead of print. PMID 41265546